CLINICAL TRIAL: NCT05325606
Title: Registry-based Stroke Research in Tunisia: Multicenter Study
Brief Title: Registry-based Stroke in Tunisia
Acronym: RAV-TUN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, A head of Emmergency Departement in Monastir, University of Monastir
Other Study IDs: Tunisia Stroke
Record Dates: First submitted 2022-03-14; First posted 2022-04-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-11

CONDITIONS: Stroke, Ischemic; Strokes Thrombotic; Stroke
Keywords: stroke; thrombolysis; Tunisia
MeSH Terms: conditions — Ischemic Stroke; Thrombotic Stroke; Stroke

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

SUMMARY:
Study the prevalence of strokes in the emergency department (ED) and their possible eligibility for thrombolysis.

DETAILED DESCRIPTION:
The diagnosis and management of strokes represent a great emergency that requires multidisciplinary teams and an organization of the care chain from the collection of patients at the site of the stroke to follow-up care.

That is why it is necessary to identify the prevalence of stroke in the ED in Tunisia and to evaluate their eligibility for thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

* All patients with stroke symptoms.

Exclusion Criteria:

* Refusal of inclusion

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with stroke symptoms and accept to enroll the study .
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Stroke prevalence | 1day
  After entering the ED , the patient will have a radiological and biological screening to establish his right diagnostic and then we have stroke prevalence in the ED.
Modified Rankin Scale (MRS) score change | After a month , six month , 1 year
  After discharge from ED, patients were called back in order to know information about the quality of life and the search for persistent complications.

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Professor, Principal Investigator — University of Monastir
Locations (1):
- Nouira Semir, Monastir, Tunisia